CLINICAL TRIAL: NCT06495879
Title: Study of The Association Between Triglyceride Glucose Index and Severity of Coronary Artery Disease
Brief Title: Association Between Triglyceride Glucose Index and Severity of Coronary Artery Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fatma Mohamed Abdelaal, Fatma Mohamed Abdelal, Sohag University
Other Study IDs: Soh-Med-24-06-02MS
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronary artery disease (CAD) is a chronic cardiovascular disease occurring due to atherosclerotic occlusion of the coronary arteries (1).

Acute coronary syndrome (ACS) is the most severe type of Coronary artery disease including unstable angina(UA) , St -elevation myocardial infarction (STEMI) Non ST elevation mayocardial infarction (NSTEMI) (2).

Despite the use of current guidline-recommended therapeutics including Percutaneous coronary intervention (PCI) or coronary Artery bypass Grafting (CABG) and optimal drug treatments some patients with ischemic heart disease (IHD) remain at high risk for recurrent Cardio vascular events(3).

Triglyceride glucose index (TYG) has a good potential in predicting poor cardiovascular prognosis in patients with IHD (4).

ELIGIBILITY:
Inclusion Criteria:

- This study will be conducted on patients investigated for IHD by coronary angiography at coronary catheterization unit at sohag university hospital

Exclusion Criteria:

* 1- Patients younger than 18 years. 2- Patients with malignant tumor disease . 3- Patients with infectious or sever liver or kidney disease . 4- Patients lacked data on HbA1c,FPG,TG.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted on patients investigated for IHD by coronary angiography at coronary catheterization unit at sohag university hospital
  Exclusion Criteria:
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Triglyceride glucose index | 6 months
  Association between Triglyceride glucose index and severity of coronary artery disease

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Virani SS, Alonso A, Aparicio HJ, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Cheng S, Delling FN, Elkind MSV, Evenson KR, Ferguson JF, Gupta DK, Khan SS, Kissela BM, Knutson KL, Lee CD, Lewis TT, Liu J, Loop MS, Lutsey PL, Ma J, Mackey J, Martin SS, Matchar DB, Mussolino ME, Navaneethan SD, Perak AM, Roth GA, Samad Z, Satou GM, Schroeder EB, Shah SH, Shay CM, Stokes A, VanWagner LB, Wang NY, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2021 Update: A Report From the American Heart Association. Circulation. 2021 Feb 23;143(8):e254-e743. doi: 10.1161/CIR.0000000000000950. Epub 2021 Jan 27. PMID 33501848
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- [Background] Ray KK, Colhoun HM, Szarek M, Baccara-Dinet M, Bhatt DL, Bittner VA, Budaj AJ, Diaz R, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Loizeau V, Lopes RD, Moryusef A, Murin J, Pordy R, Ristic AD, Roe MT, Tunon J, White HD, Zeiher AM, Schwartz GG, Steg PG; ODYSSEY OUTCOMES Committees and Investigators. Effects of alirocumab on cardiovascular and metabolic outcomes after acute coronary syndrome in patients with or without diabetes: a prespecified analysis of the ODYSSEY OUTCOMES randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Aug;7(8):618-628. doi: 10.1016/S2213-8587(19)30158-5. Epub 2019 Jul 1. PMID 31272931